CLINICAL TRIAL: NCT06472297
Title: Diabetes Prevention Combining CGM and Artificial Intelligence Health Education
Brief Title: Continuous Glucose Monitoring in Prediabetes
Acronym: G1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, David S Black, PhD, Associate Professor of Population and Public Health Sciences, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UP-23-01001; P50MD017344 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pre-diabetes
Keywords: Prediabetes; Glucose management; Feedback; Narrative education; Artificial intelligence; Contingency-shaped learning
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Intervention Model Description: A case series of participants wear an unmasked CGM sensor for a condition lasting 20 days while recording daily narratives of their experience.
Masking Description: The CGM system feedback is unmasked. The CGM is automatically recorded and does not require an outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Unmasked CGM feedback (Experimental): The CGM system is used by the participant according to manufacturer instructions for the condition interval in their normal living environment.
  Interventions: Device: The continuous glucose monitoring system

INTERVENTIONS:
Device: The continuous glucose monitoring system — CGM device worn on back of the arm and glucose readings are shown on the participant's smartphone as a continuous data stream.
  Other Names: CGM feedback

SUMMARY:
The objective of this project is to develop a behavioral intervention that combines wearable continuous glucose monitoring (CGM) with smartphone feedback and educational video clips generated by artificial intelligence (AI) software to improve glycemic control among individuals with pre-diabetes. The goal is to prevent transition to type 2 diabetes.

DETAILED DESCRIPTION:
Video narratives will be provided by Latino community health workers, known as Promotores de Salud (PdS), who will wear and experience the continuous glucose monitoring (CGM) system and its glycemic variability feedback. Study 1 (G1) is a Phase 0 intervention development study, enrolling a sample of 20 Spanish- and/or English-speaking PdS who test positive for pre-diabetes via a finger prick screening. Participants will wear CGM devices for 20 days, during which they will record daily narratives about their experiences with the CGM feedback and their glucose variability. Structured interviews between staff and participants will explore the benefits and barriers of CGM use. These recorded video clips will serve as the foundation for educational cinematic smartphone videos for future interventions. Artificial intelligence (AI) tools will be used to translate the text, audio, and video clips into various languages for broad dissemination. Blood glucose levels in mg/dL will be recorded continuously over the wear period.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes by finger prick blood A1C%
* Centers for Disease Control and Prevention (CDC) prediabetes risk test score of 5 or higher
* Willingness to wear CGM sensor
* Latino community health worker

Exclusion Criteria:

* Currently pregnant
* Less than 18 years of age, which is adult in California
* Diagnosed with any disorder that interferes with glucose
* Influential medical disorder/event affecting ability to participate in study
* Incompatible smartphone device not pairing with Dexcom G6 app

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Black, PhD MPH, Principal Investigator — University of Southern California
Locations (1):
- Southern California Center for Latino Health SCCLH, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing is set up with affiliate P50 Center universities and hospitals under a registered data use agreement (DUA). Data will be posted on the Open Science Framework url
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Researchers can obtain de-identified data and statistical codes after publication of the study outcomes by email request and as supplemental material in future journal publications.
Access Criteria: Request from author or see study publication supplemental material on the journal website.
URL: https://www.usc.edu

REFERENCES:
- See also: Dexcom G CGM system specifications — https://www.dexcom.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and preliminary screening activities occurred between 5/24/2024 and 8/30/2024, using baseline screening telephone calls. The Study Start Date of 6/1/2024 reflects the date on which the first participant was formally enrolled in the study. The target population included 20 community health workers who had been actively working within the past six months, were diagnosed with prediabetes, and primarily resided in Los Angeles County.
Groups:
- Unmasked CGM Feedback (Single Study Arm): The CGM system is used by the participant according to manufacturer instructions for the condition interval in their normal living environment.
  The continuous glucose monitoring system: CGM device worn on back of the arm and glucose readings are shown on the participant's smartphone as a continuous data stream.
Period: Overall Study
Arm/Group | Unmasked CGM Feedback (Single Study Arm)
Started | 23
Completed | 21 (2 withdrew prior to protocol completion)
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Baseline measures were collected and reported for all 23 enrolled participants. Primary outcome analyses were conducted participants with sufficient continuous glucose monitoring data (≥2 days of valid data per 10-day period), as pre-specified for the two-timepoint design.
Arm/Group | Unmasked CGM Feedback (Single Study Arm)
Number analyzed (Participants) | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.0 [45.5 to 56.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 20
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
Highest level of education [Count of Participants; unit: Participants]
  High School or Less | 11
  Some College or Vocational Training | 1
  College Degree or Higher | 11
Current employment status [Count of Participants; unit: Participants]
  Employed | 18
  Unemployed | 1
  Retired | 2
  Homemaker | 2
  Student | 0
Total household income [Count of Participants; unit: Participants]
  Less than $10,000 | 2
  $10,000 to $29,999 | 7
  $30,000 to $49,999 | 9
  $50,000 to $69,999 | 3
  $70,000 to $89,999 | 1
  $90,000 to $149,999 | 1
  $150,000 or more | 0
Health insurance [Count of Participants; unit: Participants]
  Public | 17
  Private | 5
  Self-cash paying | 1
Centers for Disease Control and Prevention (CDC) prediabetes risk score [Count of Participants; unit: Participants] — The CDC Prediabetes Risk Score is a questionnaire-based score calculated from age, sex, family history, gestational diabetes history, hypertension, physical activity, and weight category. Higher scores indicate greater diabetes risk (worse outcomes), while lower scores indicate lower risk (better outcomes). A score of 5 or higher indicates increased risk for having prediabetes and are at high risk for type 2 diabetes.
  Participants
    Scored under 5 | 4
    Scored 5 or higher | 19
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m²] | 31.8 [29.0 to 36.6]
Physical Activity Level (International Physical Activity Questionnaire [IPAQ]) [Count of Participants; unit: Participants] — IPAQ is a validated self-report instrument designed to estimate physical activity over the previous 7 days. Participants reported the frequency (days per week) and duration (minutes per day) of walking, moderate-intensity activity, and vigorous-intensity activity.
  Total physical activity was calculated in metabolic equivalent task minutes per week (MET-min/week). Based on total MET-min/week, participants were categorized into low, moderate, or high physical activity levels, according to established IPAQ criteria.
  Participants
    Low | 6
    Moderate | 7
    High | 10
HbA1c (%) [Count of Participants; unit: Participants] — Finger prick HbA1c (%)
  Participants
    HbA1c < 5.7% | 11
    HbA1c ≥ 5.7% | 12
Self-reported history of prediabetes [Count of Participants; unit: Participants]
  Yes | 14
  No | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Glucose (mg/dL) From Baseline
Description: Mean glucose was derived from continuous glucose monitoring (CGM) data obtained from the Dexcom Clarity system. Raw glucose values were processed and analyzed using the R statistical software package iglu to generate the full CGM variability metrics panel. For each participant, mean glucose was calculated separately for each 10-day assessment period. The outcome measure represents the change in mean glucose, defined as the difference between the baseline (Phase A) 10-day assessment period and the subsequent (Phase B) 10-day assessment period.
Time Frame: Up to 20 days of continuous CGM wear, comprising two sequential 10-day assessment periods (baseline Phase A and subsequent Phase B).
Population: Participants included in the analysis had sufficient continuous glucose monitoring (CGM) data. Inclusion required at least 2 days of valid CGM data within each 10-day assessment period. Three participants were excluded: two withdrew before completion of data collection, and one was later deemed ineligible based on protocol criteria identified after enrollment. Primary outcome analyses were therefore conducted on 20 participants.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Unmasked CGM Feedback (Single Study Arm)
Number analyzed (Participants) | 20
mg/dL | 2.1 [-7.4 to 9.3]
Statistical Analysis 1: Comparison: Unmasked CGM Feedback (Single Study Arm); Test type: Other — Single group; p = 0.8, Wilcoxon Signed Rank test — A two-sided significance level of 0.05 was used. No adjustment for multiple comparisons was required due to a single primary outcome; The Wilcoxon signed-rank test was used to compare paired within-participant mean glucose values between Phase A and Phase B; Median Difference (Net) = 2.1 — The median difference represents the median change in mean glucose between Phase A and Phase B

2. Other Pre Specified Outcome: Total Duration of Participant-Generated Narrative Video Recordings
Description: Total duration, in minutes, of narrative video recordings generated by participants, including daily selfie-style reflections recorded during the continuous glucose monitor (CGM) wear period and post-study interview recordings (as a measure of feasibility).
  The total number of minutes of recorded narrative video content was calculated by summing the duration of all daily reflection videos and post-study interview recordings across participants. Results are reported as total minutes.
Time Frame: Up to 20 days during the CGM wear period, plus post-study interview recordings.
Population: All participants that provided at least 1 video.
Measure: Number; unit: minutes
Arm/Group | Unmasked CGM Feedback (Single Study Arm)
Number analyzed (Participants) | 21
minutes | 723

ADVERSE EVENTS:
Time Frame: From participant enrollment through end of study follow-up (20 days)
Arm/Group | Unmasked CGM Feedback (Single Study Arm)
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Unmasked CGM Feedback (Single Study Arm) (N=23)
Sensor site pain (Skin and subcutaneous tissue disorders) | 3 — Localized pain at the site of sensor placement.
Sensor site itching (Skin and subcutaneous tissue disorders) | 1 — Itchiness at the sensor adhesive site reported by the participant; resolved without intervention and without associated redness or inflammation.

LIMITATIONS AND CAVEATS:
The Phase 0 intervention goal raises few concerns regarding scientific rigor; however, focusing on a single major racial/ethnic group limits the generalizability of the content to other racial/ethnic groups, which will be addressed in future work.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT06472297/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT06472297/SAP_001.pdf